CLINICAL TRIAL: NCT01225224
Title: Phase I Study of ASP015K: Single-Dose and Multiple-Dose Oral Administration in Healthy Nonelderly Men
Brief Title: Single and Multiple Oral Administration Study of ASP015K in Healthy Nonelderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 015K-CL-HV03
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2019-09

CONDITIONS: Pharmacokinetics of ASP015K; Healthy Volunteer
Keywords: ASP015K; Ethnic difference
MeSH Terms: interventions — peficitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- ASP015K Single Japanese Group (Experimental): Participants will be administered a single dose of ASP015K in three stages, each stage corresponding to a different dosage level.
  Interventions: Drug: peficitinib
- ASP015K Single Caucasian Group (Experimental): Participants will be administered a single dose of ASP015K in three stages, each stage corresponding to a different dosage level.
  Interventions: Drug: peficitinib
- Placebo Single Japanese Group (Placebo Comparator): Participants will be administered a single dose of placebo in three stages, each stage corresponding to a different dosage level.
  Interventions: Drug: Placebo
- Placebo Single Caucasian Group (Placebo Comparator): Participants will be administered a single dose of placebo in three stages, each stage corresponding to a different dosage level.
  Interventions: Drug: Placebo
- ASP015K Multiple Group (Experimental): Participants will receive ASP015K in three stages, each stage corresponding to a different dosage level. ASP015K will be administered at 12-hour intervals after breakfast and dinner for seven days.
  Interventions: Drug: peficitinib
- Placebo Multiple Group (Placebo Comparator): Participants will receive placebo in three stages, each stage corresponding to a different dosage level. Placebo will be administered at 12-hour intervals after breakfast and dinner for seven days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
  Arms: ASP015K Multiple Group; ASP015K Single Caucasian Group; ASP015K Single Japanese Group
Drug: Placebo — oral
  Arms: Placebo Multiple Group; Placebo Single Caucasian Group; Placebo Single Japanese Group

SUMMARY:
A study to evaluate the safety, tolerability and PK profiles of single and multiple doses of ASP015K in healthy nonelderly men.

DETAILED DESCRIPTION:
This study consists of two parts; single and multiple administration parts. In single administration part, multiple dose levels of ASP015K or placebo are administered to Japanese and Caucasian men to evaluate whether there is ethnic differences in the pharmacokinetics and pharmacodynamics of ASK015K. In multiple administration part, drugs are administered only to Japanese volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy judged by the investigator or subinvestigator on the basis of physical examination and all test results
* Weight

  * Japanese: ≥ 50.0 kg to < 80.0 kg
  * Caucasians: ≥ 50.0 kg to < 100.0 kg
* BMI

  * Japanese: ≥ 17.6 kg/m2 to < 26.4 kg/m2
  * Caucasians: ≥ 18.0 kg/m2 to < 30.0 kg/m2
* Written informed consent obtained from the subject personally

Exclusion Criteria:

* Administered drug in another clinical study or a post-market clinical study in the 120 days prior to the study
* Collection of 400 mL of whole blood within 90 days prior to the study,

  200 mL of whole blood within 30 days prior to the study or blood components within 14 days prior to the study
* Received or is scheduled to receive drug treatment within 7 days prior to the drug administration
* A history of drug allergies
* Upper gastrointestinal symptoms, e.g., nausea, vomiting or stomachache, within 7 days prior to the drug admission
* Concurrent or previous liver disease, e.g., viral hepatitis or drug-induced hepatic injury
* Concurrent or previous heart disease, e.g., congestive heart failure, angina pectoris or arrhythmias requiring treatment
* Concurrent or previous kidney disease, e.g., acute renal failure,

glomerulonephritis or interstitial nephritis (except for previous urinary

calculus)

* Concurrent or previous cerebrovascular disease, e.g., cerebral infarction
* Concurrent or previous malignancy
* Concurrent or previous active or recurrent infection, e.g., hepatitis B,

hepatitis C or syphilis

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11-18 (Actual); Primary Completion 2010-03-10 (Actual); Study Completion 2010-03-10 (Actual)

PRIMARY OUTCOMES:
Safety evaluated by the incidence of AE, vital signs , standard 12-lead ECG and Laboratory tests | For 48 hours after administration

SECONDARY OUTCOMES:
Plasma unchanged drug concentration | For 48 hours after administration
Urinary unchanged drug concentration | For 48 hours after administration
Transcription factor phosphorylation level | For 48 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kyushu, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Shibata M, Hatta T, Saito M, Toyoshima J, Kaneko Y, Oda K, Nishimura T. Pharmacokinetics, Pharmacodynamics, and Safety of Peficitinib (ASP015K) in Healthy Male Caucasian and Japanese Subjects. Clin Drug Investig. 2020 May;40(5):469-484. doi: 10.1007/s40261-020-00910-w. PMID 32274653